CLINICAL TRIAL: NCT01850004
Title: Open-Label Single Arm Phase 2 Study Evaluating Dasatinib Therapy Discontinuation In Patients With Chronic Phase Chronic Myeloid Leukemia (CP-CML) With Stable Complete Molecular Response (CMR) DASFREE
Brief Title: Open-Label Study Evaluating Dasatinib Therapy Discontinuation in Patients With Chronic Phase Chronic Myeloid Leukemia With Stable Complete Molecular Response
Acronym: DASFREE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: ICON plc (Industry); PPD Development, LP (Industry); Molecular MD (Unknown); European Organisation for Research and Treatment of Cancer - EORTC (Network); MultiPharma (Unknown); Steering Committee (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CA180-406; 2012-001421-27 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-09 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib (Experimental): Dasatinib 50, 80, 100, 140, 180 mg tablets by mouth, once daily, up to 60 months
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib
  Other Names: Sprycel

SUMMARY:
The study purpose is to test the hypothesis that Chronic Phase Chronic Myeloid Leukemia (CP-CML) patients with stable Complete Molecular Response (CMR) who discontinue Dasatinib treatment are able to maintain a sustained remission in the long-term, with undetectable or minimally detectable BCR-ABL residual disease.

DETAILED DESCRIPTION:
Primary Purpose: Protocol designed to evaluate remission of disease after treatment discontinuation. Treatment re-started if relapse occurs

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria

* Signed Written Informed Consent
* Target Population

  1. Men and women diagnosed with CP-CML, on treatment with dasatinib for a minimum of 2 years at the time of enrollment and in dasatinib-induced complete molecular remission ongoing for at least 1 year prior to study entry.
  2. Patients are eligible if they have been in stable dasatinib induced CMR for a minimum of nine months, documented by at least three assessments, conducted 2 - 6.5 months apart, at a local lab.
  3. Subjects who have received dasatinib beyond first or second line treatment and meet other enrollment criteria are eligible for the study provided prior Tyrosine-kinase inhibitors (TKI) were discontinued due to intolerance or lack efficacy, although only one instance of lack of efficacy to TKI is allowed.
  4. Eastern Co-Operative Group (ECOG) Performance Status (PS) of 0-1
* Age and Reproductive Status

  1. Men and women, ages ≥18
  2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the restart of study drug
  3. Women must not be breastfeeding
  4. WOCBP must agree to follow instructions for method(s) of contraception at the restart of treatment with study drug (dasatinib) and for the duration treatment plus 30 days (duration of ovulatory cycle) for a total of 30 days post-treatment completion
  5. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for 90 days after study entry (withdrawal of dasatinib), at restart of study drug (dasatinib) and for the duration of treatment with study drug (dasatinib) plus 90 days (duration of sperm turnover) for a total of 90 days post-treatment completion

Exclusion Criteria:

* Target Disease Exceptions

  1. Patients who have not achieved a 1-log reduction in BCR-ABL transcript levels compared with baseline as determined by local standards or > 10% IS [International Standard]) documented at 3.0-6.5 months since the initial start of dasatinib therapy.
  2. Patients who have previously undergone hematopoietic stem cell transplantation (SCT) or who are scheduled for SCT
  3. Previous diagnosis of CML accelerated phase or blast crisis
* Medical History and Concurrent Diseases

  1. Prior or concurrent malignancy, except the following:

     * Curatively treated basal cell or squamous cell skin cancer
     * Cervical carcinoma in situ
     * Adequately treated Stage I or II cancer from which the subject is currently in complete remission
     * Any other cancer from which the subject has been disease free for 3 years
  2. A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy in case re-initiation of dasatinib is needed.
  3. Uncontrolled or significant cardiovascular disease
  4. Subjects with prior history of pericardial effusion or pleural effusion that required thoracentesis are excluded. Subjects with prior history of pericardial or pleural effusion that was clinically manageable and a maintained CMR for ≥ 1 year on a stable dose of dasatinib are allowed.
  5. History of significant bleeding disorder unrelated to CML
* Allergies and Adverse Drug Reaction

  a. Subjects with known hypersensitivity to excipients of Dasatinib tablets
* Sex and Reproductive Status

  1. Patients who are pregnant or breastfeeding or likely to become pregnant
  2. Men whose partner is unwilling or unable to avoid pregnancy
* Other Exclusion Criteria

  1. Patients with a history of non-compliance to CML treatment and monitoring requirements
  2. Prisoners or subjects who are involuntarily incarcerated
* Additional Criteria for Patients Eligible to Restart Dasatinib

  * Any patient who has lost MMR and is eligible for re-starting dasatinib therapy must not have developed a condition that precludes dasatinib use.

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (28):
- United States (8):
  - Local Institution - 0006, Duarte, California
  - Local Institution - 0029, Los Angeles, California
  - Local Institution - 0001, San Franisco, California
  - Local Institution - 0013, Chicago, Illinois
  - Local Institution - 0024, Hackensack, New Jersey
  - Local Institution - 0028, New York, New York
  - Local Institution - 0011, Dallas, Texas
  - Local Institution - 0023, Houston, Texas
- Local Institution - 0005, Toronto, Ontario, Canada
- France (4):
  - Local Institution - 0012, Paris
  - Local Institution - 0003, Pessac
  - Local Institution - 0030, Pierre-Bénite
  - Local Institution - 0002, Vandœuvre-lès-Nancy
- Germany (5):
  - Local Institution - 0019, Rostock, Mecklenburg-Vorpommern
  - Local Institution - 0026, Aachen
  - Local Institution - 0020, Berlin
  - Local Institution - 0021, Mannheim
  - Local Institution - 0022, Ulm
- Italy (6):
  - Local Institution - 0025, Catania
  - Local Institution - 0017, Florence
  - Local Institution - 0027, Napoli
  - Local Institution - 0015, Orbassano
  - Local Institution - 0018, Roma
  - Local Institution - 0016, Rome
- Spain (4):
  - Local Institution - 0014, Oviedo, Principality of Asturias
  - Local Institution - 0009, Las Palmas de Gran Canaria
  - Local Institution - 0010, Madrid
  - Local Institution - 0008, Málaga

REFERENCES:
- [Derived] Shah NP, Garcia-Gutierrez V, Jimenez-Velasco A, Larson SM, Saussele S, Rea D, Mahon FX, Levy MY, Gomez-Casares MT, Mauro MJ, Sy O, Martin-Regueira P, Lipton JH. Treatment-free remission after dasatinib in patients with chronic myeloid leukaemia in chronic phase with deep molecular response: Final 5-year analysis of DASFREE. Br J Haematol. 2023 Sep;202(5):942-952. doi: 10.1111/bjh.18883. Epub 2023 May 29. PMID 37246588
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Total: Prior to study entry participants received dasatinib as treatment for a minimum of 2 years. Upon enrollment dasatinib will be discontinued. Dasatinib will be restarted if major molecular response is lost during the off-treatment period at the dose level received before study entry. The participant will remain on treatment for the duration of the study.
Period: Overall Study
Arm/Group | Total
Started | 84
Restart Treatment (Restarted treatment due to failure to maintain MMR levels of BCL-ABL) | 47
Discontinued Study Treatment After Restart | 47
Completed (Completed study) | 60
Not Completed | 24
Not completed — Poor/Non-compliance | 1
Not completed — Participant Withdrew Consent | 9
Not completed — Participant Request to Discontinue Treatment | 2
Not completed — Adverse Event Unrelated to Study Drug | 1
Not completed — Adverse Event Related to Study Drug | 4
Not completed — Other Reasons | 2
Not completed — Participant No Longer Meets Study Criteria | 1
Not completed — Maximum Clinical Benefit | 4

BASELINE CHARACTERISTICS:
Arm/Group | Total
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 75
  Black/African American | 3
  Asian | 1
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Major Molecular Response (MMR) Rate
Description: Major Molecular Response (MMR) rate at 12 months is the percentage of participants who maintain MMR (BCR-ABL transcripts < 0.1% on the International Scale [IS]) at 12 months after Dasatinib discontinuation without restarting Dasatinib
Time Frame: At 12 months after Dasatinib discontinuation (assessed up to approximately June 4, 2018)
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Total
Number analyzed (Participants) | 84
Percentage of Participants | 47.6 [36.6 to 58.8]

2. Secondary Outcome: Event-Free Survival (EFS) Rate
Description: Event-free survival (EFS) rate is defined as the percentage of surviving participants with no loss of Major Molecular Response (MMR) at the specified timepoints after dasatinib discontinuation. MMR is defined as BCR-ABL transcripts < 0.1% IS. Loss of MMR is defined per the European LeukemiaNet (ELN) definition of progression. Progression is defined as Transformation to Accelerated Phase or Blast Crisis (AP/BC):
  Accelerated Phase (AP) Blasts in PB or BM 15-29%; Blast + promyelocytes ≥ 30% with blasts < 30% or ACA in Ph+ cells (clonal progression), or basophils in blood ≥ 20%,or platelets < 100 x 10^9 /L unrelated to therapy
  Blastic Phase or Crisis (BP/BC) Blasts in PB or BM ≥ 30%, or extramedullary blast cell involvement (with exception of spleen and liver)
  The date of progression is defined as the date any of the above criteria is first met. Participants who have not progressed will be censored on the date of last examination.
Time Frame: From 12 months after Dasatinib treatment discontinuation to every 12 months thereafter (up to approximately 60 months)
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Total
Number analyzed (Participants) | 84
Percentage of participants
  At 12 months | 48.7 [38.0 to 59.4]
  At 24 months | 46.3 [35.6 to 57.0]
  At 36 months | 45.0 [34.3 to 55.7]
  At 48 months | 43.8 [33.1 to 54.4]
  At 60 months | 43.8 [33.1 to 54.4]

3. Secondary Outcome: Relapse-Free Survival (RFS) Rate
Description: RFS is the percentage of participants who did not relapse at the specified timepoints. Participants who did not relapse were censored on the date of their last molecular assessment. Relapse is defined as any of the following events while on study: the loss of Major Molecular Response (MMR), loss of Complete Cytogenetic Response (CCyR), loss of Complete Hematologic Response (CHR) or progression to advanced/blastic phase.
  MMR is defined as BCR-ABL transcripts < 0.1% IS. Cytogenetic response (CyR) is based on the prevalence of Ph+ cells in metaphase from bone marrow (BM) sample based on evaluation of at least 20 metaphases. CCyR is defined as 0% Ph+ cells in metaphase in BM. CHR is obtained when all the following criteria are met in peripheral blood (PB) sampling: white blood cell ≤10,000/mm3; Platelets < 450,000/mm3; PB basophils <5%; No blasts or promyelocytes in PB; <5% myelocytes plus metamyelocytes in PB; No extramedullary involvement (including no hepatomegaly or splenomegaly).
Time Frame: From 12 months after Dasatinib treatment discontinuation to every 6 months thereafter (up to approximately 60 months)
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Total
Number analyzed (Participants) | 84
Percentage of Participants
  At 6 Months | 61.9 [51.5 to 72.3]
  At 12 Months | 48.7 [38.0 to 59.4]
  At 18 Months | 47.5 [36.8 to 58.2]
  At 24 months | 46.3 [35.6 to 57.0]
  At 30 months | 46.3 [35.6 to 57.0]
  At 36 months | 45.0 [34.4 to 55.7]
  At 42 months | 43.8 [33.1 to 54.4]
  At 48 months | 43.8 [33.1 to 54.4]
  At 54 months | 43.8 [33.1 to 54.4]
  At 60 months | 43.8 [33.1 to 54.4]

4. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: Progression free survival (PFS) is defined as the percentage of participants who experienced death (due to any cause) or accelerated phase, or blast crisis. Participants who neither progress nor die will be censored on the date of their last molecular assessment. Progression is defined as Transformation to Accelerated Phase or Blast Crisis (AP/BC) Accelerated Phase (AP) Blasts in PB or BM 15-29%; Blast + promyelocytes >= 30% with blasts < 30% or ACA in Ph+ cells (clonal progression), or basophils in blood >= 20%,or platelets < 100 x 109 /L unrelated to therapy Blastic Phase or Crisis (BP/BC) Blasts in PB or BM >= 30%, or extramedullary blast cell involvement (with the exception of spleen and liver)
Time Frame: From 12 months after Dasatinib treatment discontinuation to every 6 months thereafter (up to approximately 60 months)
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Total
Number analyzed (Participants) | 84
Percentage of participants
  At 6 months | 100.0 [100.0 to 100.0]
  At 12 months | 100.0 [100.0 to 100.0]
  At 18 months | 100.0 [100.0 to 100.0]
  At 24 months | 98.7 [96.2 to 100.0]
  At 30 months | 98.7 [96.2 to 100.0]
  At 36 months | 98.7 [96.2 to 100.0]
  At 42 months | 98.7 [96.2 to 100.0]
  At 48 months | 98.7 [96.2 to 100.0]
  At 54 months | 98.7 [96.2 to 100.0]
  At 60 months | 98.7 [96.2 to 100.0]

5. Secondary Outcome: Number of Participants Who Experience Intermittent Loss of Complete Molecular Response (CMR) (MR4.5) But no Loss of Major Molecular Response (MMR)
Description: The number of participants who did not lose major molecular response (MMR) 60 months after discontinuing study treatment who were in MR4.5 at the time of discontinuation and lost MR4.5. Molecular response will be assessed using BCR-ABL transcript levels measurement by real-time quantitative polymerase chain reaction (Q-PCR). MMR is defined as BCR-ABL transcripts < 0.1% Internal Standard (IS). CMR (MR4.5) defined as ≤ 0.0032% (IS) or ≥ 4.5 log reduction of BCR-ABL transcript levels molecular response.
Time Frame: 60 months after last dose
Population: Participants with no loss of major molecular response (MMR)
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 31
Participants | 19

6. Secondary Outcome: Number of Participants Who Did Not Experience Loss of Complete Molecular Response (CMR) (MR4.5) and Major Molecular Response (MMR)
Description: Assessment of BCR-ABL kinetics in patients who are in CMR (MR4.5) or less when transcript levels are still measurable. CMR (MR4.5) defined as ≤ 0.0032% (IS) or ≥ 4.5 log reduction of BCR-ABL transcript levels molecular response.
Time Frame: From 12 months after Dasatinib treatment discontinuation to 5 years after the first visit of the last enrolled participant (up to approximately 82 months)
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 31
Participants | 12

7. Secondary Outcome: Time to Transformation to Accelerated Phase/Blast Crisis (AP/BC)
Description: Time to Transformation to AP/BC is defined as the rate at which participants experienced transformation to accelerated phase/blast crisis (AP/BC) since discontinuation. Participants who did not develop to AP, late phase, or BC phase were censored on their last molecular measurement date.
Time Frame: as for outcome 6
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total
Number analyzed (Participants) | 84
Months | NA [NA to NA] — The median, lower and upper limits were incalculable due to insufficient number of events

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from dasatinib treatment discontinuation to the date of death (due to any cause) or last known alive date. Participants who do not die will be censored on their last known alive date.
Time Frame: From 12 months after Dasatinib treatment discontinuation to the date of death or last known alive date (up to approximately 82 months)
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total
Number analyzed (Participants) | 84
Months | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events.

9. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the time from treatment discontinuation to the date of progression or death (due to any cause), whichever occurs first. Participants who neither progress nor die will be censored on the date of their last molecular assessment.
Time Frame: From treatment discontinuation to the date of progression or death due to any cause, whichever occurs first (up to 82 months)
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total
Number analyzed (Participants) | 84
Months | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events.

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their enrollment to study completion, (up to approximately 87 months). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 85 months)
Description: The number at Risk for All-Cause Mortality represents all enrolled Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication during re-treatment.
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 1/84
Serious Adverse Events (participants affected / at risk) | 8/47
Other Adverse Events (participants affected / at risk) | 42/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=47)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
External ear cellulitis (Infections and infestations) | 1
Polychondritis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=47)
Neutropenia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 5
Fatigue (General disorders) | 10
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 4
Nasopharyngitis (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Viral infection (Infections and infestations) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 6
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT01850004/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT01850004/SAP_001.pdf